CLINICAL TRIAL: NCT03856268
Title: Understanding the Roles of Estradiol and Follicle-stimulating Hormone in Adipocyte Remodeling Following Surgical and Pharmacology-induced Menopause (RESUME-2 Study)
Brief Title: Understanding the Roles of Hormones in Adipocyte Remodeling Following Menopause
Acronym: RESUME-2
Status: Withdrawn | Type: Observational
Why Stopped: PI left the institution.
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: University of Colorado, Denver (Other); University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Kara Marlatt, Postdoctoral Researcher - John S McIlhenny Skeletal Muscle Physiology - Ravussin, Pennington Biomedical Research Center
Other Study IDs: PBRC 2019-010
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Menopause Surgical; Estrogen Deficiency; Adiposity; Follicle-Stimulating Hormone Deficiency; Hormone Deficiency
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Adipose tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ARM 1: 'Surgical Menopause' Group: Premenopausal women having an oophorectomy.
  Interventions: Procedure: 'Surgical Menopause' Group
- ARM 2: "Drug-Induced Menopause': Premenopausal women with gonadal suppression
  Interventions: Drug: 'Drug-Induced Menopause' Group
- 'Comparative (Control)' Group: Premenopausal women with regular cycles.

INTERVENTIONS:
Procedure: 'Surgical Menopause' Group — Women undergoing laparoscopic oophorectomy surgery ('surgical menopause') will be enrolled at Pennington Biomedical.
  Other Names: 'Bilateral Oophorectomy Surgery' Group
  Groups: ARM 1: 'Surgical Menopause' Group
Drug: 'Drug-Induced Menopause' Group — Women undergoing gonadal suppression via leuprolide acetate (Lupron [AbbVie Inc.]) will be enrolled at the University of Colorado-Denver.
  Other Names: 'Pharmacology-Induced Menopause' Group
  Groups: ARM 2: "Drug-Induced Menopause'

SUMMARY:
The overarching aims of this study are to:

1. Characterize the rate of in vivo adipogenesis, and changes in adipose tissue gene and protein expression, in the scABD and scFEM depots of women undergoing surgical menopause (↓E2, ↑FSH).
2. Characterize the rate of in vivo adipogenesis, and changes in adipose tissue gene and protein expression, in the scABD and scFEM depots of women undergoing gonadal suppression (↓E2, ↓FSH).

DETAILED DESCRIPTION:
This is a cross-sectional study where two groups of premenopausal women (ages 18-50 y) will be enrolled in a parallel arm study:

* Arm 1 (Surgical Menopause): up to 6 women undergoing laparoscopic, elective bilateral oophorectomy [Site: Pennington Biomedical Research Center].
* Arm 2 (Pharmacology-Induced Menopause): up to 6 women undergoing gonadal suppression via leuprolide acetate (Lupron [AbbVie Inc.]) [Site: UC-Denver].

We will compare each arm of women to non-oophorectomized, premenopausal women (controls) with normal menstrual cycles (Apple&Pear study; NCT01748994; PI: Ravussin) selectively matched (1:2) for age and BMI. The Apple&Pear study uses the same in vivo adipogenesis labeling protocol, with similar age and BMI criteria, as the proposed study.

ELIGIBILITY:
INCLUSION CRITERIA:

* Healthy female
* Ages 18-50 y
* Planning to have either a laparoscopic bilateral oophorectomy or a laparoscopic unilateral oophorectomy (which would result in no remaining ovaries)
* Are willing to drink heavy water (2H2O) over an 8-week period
* Medically cleared for participation in the study by OB/GYN and Medical Investigator
* Are willing to have blood and fat tissue stored for future use

EXCLUSION CRITERIA:

* Meet either of the following criteria:
* Have all 3 of the major menopause-related symptoms [hot flashes, mood swings, insomnia (trouble sleeping)]
* Have 2 of the major menopause-related symptom combinations [hot flashes and mood swings, or hot flashes and insomnia (trouble sleeping)]
* Unstable weight in the last 3 months [gain or loss >7 lb (or 3.2 kg)]
* History of clinically diagnosed diabetes or a fasting blood glucose >126 mg/dL
* Chronic use of systemic glucocorticoids, antipsychotic/antidepressant medications, thiazolidinediones and other medications that cause clinically significant weight gain, weight loss or are known to make changes in fat cell number/size *
* Previous bariatric surgery (or other surgeries) for obesity or weight loss (< 3 years ago)
* Use of over the counter or prescription weight loss products
* History of metabolic diseases (other than diabetes)
* History of neurological disease
* History of cardiovascular disease (or other chronic diseases)
* Pregnant, planning to become pregnant, or breastfeeding
* Use of hormone replacement therapy
* Unwilling to discontinue any form or hormonal therapy (e.g., contraceptives including birth control pills, vaginal ring, injections, implant, or skin patch; hormonal supplements, etc.) upon enrollment (after the Screening Visit).

  * Inconsistent use of medications listed above will be evaluated and left up to the discretion of the Medical Investigator to evaluate safety.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Premenopausal women planning to undergo elective, laparoscopic bilateral oophorectomy surgery OR gonadal suppression via leuprolide acetate (Lupron [AbbVie Inc.]).
Study Population: Women (aged 18-50 y) will be enrolled. Women will be pre-menopausal, not pregnant, and not using hormone therapy or have medical indication for increased cancer risk.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

PRIMARY OUTCOMES:
Rate of in vivo adipogenesis (via deuterium-enrichment of adipose tissue DNA) | Change from baseline in enrichment of DNA of adipose cells with deuterium at 8 weeks
  Deuterium from the deuterium-labeled water is incorporated into the newly-synthesized DNA of newly-formed fat cell precursor cells through cell replication. The latter carry over the label when they become fat cells through differentiation. Enzymatic digestion of the fat tissue isolates the individual cells constituting the fat tissue. Centrifugation of the cell suspension allows the separation of fat cells into a floating layer and a pellet comprised of stromal-vascular cells including the fat cell precursor cells and small fat cells. As the fat cell precursor cells and small adipocytes have the property to attach quickly to plastic surfaces of culture dishes, a brief culturing of the stromal-vascular cells sorts these cells from the remaining cells. Thus, measuring the deuterium-enrichment of DNA from plastic-adherent stromal-vascular cells indicates the rate of in vivo formation of new mature fat cells and pre-adipocytes, a process collectively termed adipogenesis.

SECONDARY OUTCOMES:
Size of adipocytes | Change from baseline in size of adipocytes at 8 weeks post-surgery
  Fat cell size will be determined using osmium fixation of the lipids and measurement of their diameter with Coulter Counter followed by calculation of fat cell volume. The mean lipid content of fat cells will be calculated by multiplying the fat cell volume by the density of triolein (0.915).
Number of adipocytes | Change from baseline in number of adipocytes at 8 weeks post-surgery
  Fat cell number will be estimated by dividing the volume of adipose tissue depot of interest to the mean fat cell volume or the fat mass of the depot to the mean lipid content in fat cell.
Body composition (by Dual-energy X-ray Absorptiometry (DXA)) | Change from baseline in body composition at 8 weeks post-surgery
  Fat mass, fat-free mass, and percent body fat will be assessed using a whole-body scanner GE iDXA.
Adipose tissue gene and protein expression | Changes from baseline in gene and protein expression at 8 weeks post-surgery
  Expression levels of genes and proteins involved in adipocyte expansion and function (ERα, PPARγ2, C/EBPα, aromatase, adiponectin, and LPL), extracellular matrix remodeling and fibrosis (COL6(a1, a2, a3), COL4a1, and TGFβ), and inflammation (IL-6 and TNFα) will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Kara L Marlatt, PhD, MPH, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available upon request.